CLINICAL TRIAL: NCT02284529
Title: Evaluate the Safety of Combination of Orectalip® (Oxaliplatin), Fluorouracil and Leucovorin as Adjuvant Treatment for High-risk Stage-Ⅱ Colorectal Cancer
Brief Title: Safety of Orectalip® (Oxaliplatin) as Adjuvant Treatment for High-risk Stage-Ⅱ Colorectal Cancer
Acronym: Oxaliplatin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinphar Pharmaceutical Co., Ltd (Other)
Collaborators: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Douglas Shr-Wei Chen, Taichung Veterans General Hospital, Sinphar Pharmaceutical Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SF12099
Record Dates: First submitted 2014-10-23; First posted 2014-11-06 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-10

CONDITIONS: Stage-Ⅱ Colorectal Cancer
Keywords: high-risk stage-Ⅱ Colorectal Cancer,Orectalip,oxaliplatin
MeSH Terms: interventions — Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Orectalip® (Oxaliplatin) (Experimental): High-risk Stage-Ⅱ Colorectal Cancer treatment with Oxaliplatin 85mg/m2 in D5W 250 ml IV drip 2hrs on D1, Leucovorin 100mg/m2 in N/S 100ml IV drip 2hrs on D1, follow by 5-FU 2400mg/m2 IV infusion 24hrs on D1 to execute 8~12 cycles
  Interventions: Drug: Orectalip

INTERVENTIONS:
Drug: Orectalip — Oxaliplatin 85mg/m2 in D5W 250 ml IV drip 2hrs on D1, Leucovorin 100mg/m2 in N/S 100ml IV drip 2hrs on D1, follow by 5-FU 2400mg/m2 IV infusion 24hrs on D1
  Other Names: Fluorouracil; Leucovorin

SUMMARY:
Open- Label, Single Arm Study. To evaluate the safety profile of Orectalip® (oxaliplatin), fluorouracil and leucovorin as adjuvant therapy in the treatment of high-risk stage-Ⅱ colorectal cancer.

Primary end point:To evaluate the incidence of grade 0-3 neurosensory symptoms (paresthesia) in the end of study.

Other end points:The incidence of Grade 3 or 4 neutropenia, thrombocytopenia, anemia, nausea, diarrhea vomiting over the 12 weeks.

Safety will be evaluated including vital signs are recorded at all visits.

DETAILED DESCRIPTION:
There were 18 out of 20 patients who completed the trial and eligible for statistical analysis, 2 patients withdraw because the wound infection. There were 11 (61%) male patients and 7 (39%) female patients. The patients aged from 30 to 73 years and their mean age was 50.4 years.

The grade of each adverse event evaluation mainly allocated in Grade 0 and Grade 1. The incidence of Grade 3 or 4 was only found for the following symptoms: leucopenia, neutropenia, and anemia. One (6%) adverse event of leucopenia occurred at visit 1 and visit 2, respectively. One (6%) adverse event of neutropenia occurs at visit 1, visit 2, and visit 3, respectively; while 2 (13%) events occurred at visit 5. One patients suffered adverse event of anemia at visit 5 and visit 6.

ELIGIBILITY:
Inclusion Criteria

1. Subject must have World Health Organization performance status score less than 1.
2. Subject must have WBC more than 4,000 cells, platelet count more than 100,000, absolute neutrophil count more than 1,500 serum bilirubin level less than1.5mg, serum creatinine level less than1.5mg

Exclusion Criteria

1. Subject who has received oxaliplatin treatment
2. Subject who has history of allergy to platinum derivates agents
3. Subject who has decompensated liver function(ALT、 AST and alkaline phosphatase more than 2.5 times of upper limit of normal range).
4. Subject has serious concomitant illness preceding the entry into the study.
5. Female subject who is pregnant or breast feeding.
6. Female subject who is going to be pregnant within 6 months during treatment.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the incidence of grade 0-3 neurosensory symptoms (paresthesia) in the end of study | 6month
  Oxaliplatin 85mg/m2 in D5W 250 ml IV drip 2hrs on D1, Leucovorin 100mg/m2 in N/S 100ml IV drip 2hrs on D1, follow by 5-FU 2400mg/m2 IV infusion 24hrs on D1(cycle/ 2 weeks)To execute 12 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Hwei-Ming Wang, Chief, Principal Investigator — vghtc.crs@gmail.com
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan